CLINICAL TRIAL: NCT03617120
Title: Ergonomic Brace Wear for Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Innovation and Technology Commission, Hong Kong (Other); The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joanne Yip, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITS/297/16
Record Dates: First submitted 2018-07-25; First posted 2018-08-06 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis brace; Conventional treatment for Adolescent Idiopathic Scoliosis; In-brace correction; Trunk listing; Vertebral rotation; Interface pressure; 3D body scanning; Surface topography; Trunk asymmetry; Quality of Life

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ergonomic Brace vs hard brace (Experimental): Ergonomic Brace is a new design of scoliosis brace, which consists of a knit bodice as base and also resin bones, paddings, straps and a pelvic belt as auxiliaries for spinal correction. The purpose of the bones is to keep the posture of patient upright. Paddings are placed at the convex regions of the spine while straps are used to input directional force onto the paddings. Pelvic belt, on the other hand, is for stabilizing the pelvis in order to achieve an effective spinal correction. The biomechanical principles for the correction of spine has considered both the frontal and sagittal planes, where the overall brace mechanism follows the Rigo classification.
  Hard brace is the brace which the participants are currently using for their ongoing conservative treatment.
  Interventions: Device: Ergonomic Brace vs hard brace

INTERVENTIONS:
Device: Ergonomic Brace vs hard brace — Visit 1:
  1. Usual check-up: standing in-brace radiograph of hard brace and doctor consultation
  2. Pressure measurement of participant wearing their hard brace
  Visit 2:
  1. Brace Questionnaire (BrQ) for hard brace; Trunk Appearance Perception Scale (TAPS)
  2. 3D body scanning (before wearing the Ergonomic Brace)
  3. Fitting of the Ergonomic Brace
  4. Pressure measurement of participant wearing the Ergonomic Brace (instant)
  5. Pressure measurement of participant wearing the Ergonomic Brace (after 2 hours)
  6. 3D body scanning (after wearing the Ergonomic Brace for 2 hours)
  7. Brace Questionnaire (BrQ) for the Ergonomic Brace
  Visit 3:
  1. Standing in-brace radiograph of the Ergonomic Brace
  2. Doctor consultation

SUMMARY:
This study assesses the effectiveness of a new scoliosis brace design for adolescent idiopathic scoliosis (AIS) patients, named Ergonomic Brace, by comparing the outcome with hard brace in terms of three aspects:

1. To assess the efficacy in spinal correction
2. To evaluate the improvement made to the body appearance of AIS subjects
3. To evaluate the impacts on the quality of life (QoL) of AIS subjects

All participants will be fitted with an Ergonomic Brace and required to wear it during the days of experiment only. The ongoing treatment with hard brace will not be substituted with the Ergonomic Brace, unless its immediate treatment effect is equivalent to hard brace and with approval from the doctor.

DETAILED DESCRIPTION:
1. To assess the efficacy in spinal correction

   The efficacy of the Ergonomic Brace refers to the magnitude of spinal correction that could be obtained for patients with AIS. The assessments in this study focus on two aspects, which are i) the in-brace correction and ii) the interface pressure. In-brace correction is used to judge the quality of bracing and also a prognostic indicator for the long-term treatment outcome. Clinical parameters such as Cobb angle, vertebral rotation and trunk listing will be measured with radiographs by a single observer. Interface pressure in this study refers to the pressure between the brace and the trunk of subject. The purpose is to assess the time response of trunk to the intervention of the Ergonomic Brace, and correlation will also be made with the extent of spinal correction.
2. To evaluate the improvement made to the body appearance of AIS subjects

   The trunk aesthetic profile of AIS subjects are being affected by spinal deformities. Surface topography of the subjects will be captured by 3D body scanner, and followed by the evaluation of body aesthetics through the trunk asymmetry scales called POTSI and ATSI index. The purpose is to compare the surface topography change before and after wearing the Ergonomic Brace.
3. To evaluate the impacts on the QoL of AIS subjects

Bracing can negatively affect the QoL of patients with AIS. The Chinese version of Brace Questionnaire (BrQ) will be adopted in this study to compare the impact of hard brace and Ergonomic Brace on the QoL of AIS subjects. Difficulties experienced by AIS subjects during bracing will be highlighted and used for future improvements in scoliosis brace design.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 or older when brace is prescribed
* Risser 0 to 2
* Primary curve angles 25° to 40°
* Female, who were either pre-menarche or less than 1 year of post-menarche
* Undergoing hard brace treatment

Exclusion Criteria:

* Low risk of curve progression
* Non-idiopathic scoliosis (e.g. congenital, neuromuscular deformities)

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Immediate in-brace correction of spinal curve | 2 hours
  Cobb angle: more than/equal to 40% correction (lumbar/thoracolumbar curve); slightly less than/close to 40% correction (thoracic curve)

SECONDARY OUTCOMES:
Immediate in-brace correction of vertebral rotation assessed by the Global Torsion Index | 2 hours
  Global torsion index: to quantify detorsion by averaging the 17 segmental rotations of thoracic and lumbar vertebrae
  * Higher index score = the average segmental rotations of the 17 vertebrae is higher;
  * Lower index score = the average segmental rotations of the 17 vertebrae is lower
  The global torsion index which result from wearing the Ergonomic Brace will be compared with which of hard brace. A higher/similar detorsion percentage as hard brace is considered satisfactory.
Immediate in-brace correction of trunk listing assessed by the plumb line method | 2 hours
  Plumb line method: to assess the coronal and sagittal balance by drawing a vertical line from the mid-point of the C7 vertebra down to the sacrum
  * Positive balance: the plumb line passes more than 2 cm in front of the posterosuperior corner of the S1 vertebral body
  * Neutral balance: the plumb line passes within 2 cm of the posterosuperior corner of the S1 vertebral body
  * Negative balance: the plumb line passes more than 2 cm behind the posterosuperior corner of the S1 vertebral body
  Measurement of trunk listing is significant in the treatment of scoliosis curve, as it is related to the trunk aesthetic profile of the subjects, and besides, sagittal balance of the spine and pelvis is correlated with the progression of scoliosis. An improvement in the coronal and sagittal balance of spine resulting from wearing the Ergonomic Brace is therefore considered satisfactory.
Improvement in trunk asymmetry assessed by the POTSI index | 0 and 6 month
  Posterior Trunk Symmetry Index (POTSI): to compare the surface topography change before and after wearing the Ergonomic Brace POTSI index: a parameter used for assessing the trunk asymmetry and deformity in the coronal plane All measurements will be performed on the 3D surface topography scans. Ideal value of POTSI is zero, meaning full asymmetry of the posterior and anterior trunk respectively.
  Normal value of POTSI should lie below 27. The performance of the Ergonomic Brace in terms of improving the trunk asymmetry of participants is considered effective when the index is scored within normal value (i.e. 0-27).
Improvement in trunk asymmetry assessed by the ATSI index | 0 and 6 month
  Anterior Trunk Symmetry Index (ASTI): to compare the surface topography change before and after wearing the Ergonomic Brace ATSI index: a parameter used for assessing the trunk asymmetry and deformity in the frontal plane All measurements will be performed on the 3D surface topography scans. Ideal value of ATSI is zero, meaning full asymmetry of the posterior and anterior trunk respectively. Normal value, on the other hand, should lie below 27 for each index. The performance of the Ergonomic Brace in terms of improving the trunk asymmetry of participants is considered effective when the index is scored within normal value (i.e. 0-27).

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Yip, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Tsim Sha Tsui, Kolwoon, Hong Kong